CLINICAL TRIAL: NCT00659906
Title: Optimizing Body Composition & Health After Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 621
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Breast Neoplasm; Osteoporosis, Postmenopausal
Keywords: randomized clinical trial; cancer survivor; bone health; body composition; signs and symptoms
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis, Postmenopausal; Signs and Symptoms | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Progressive resistance training program 3 times a week for 12 months
  Interventions: Behavioral: Resistance Exercise
- 2 (Active Comparator): Flexibility training 3 times a week for 12 months
  Interventions: Behavioral: Flexibility Training

INTERVENTIONS:
Behavioral: Resistance Exercise — 60 minute sessions 3 times a week of moderate-vigorous lower and upper body free-weight strength training plus impact training (jumps). Two of the three sessions are conducted in a supervised setting at a university fitness facility and the third session is a modified version of the exercise program performed at home. Participants are in the exercise program for 12 months
  Arms: 1
Behavioral: Flexibility Training — 60 minute session 3 times a week focusing on whole body flexibility (stretching) and relaxation (progressive neuromuscular relaxation, focused breathing) exercises. Exercises are selected to be non-weight bearing and require minimal muscle strength in order to provide a contrast to the intervention arm. Two sessions are conducted in a supervised setting at a university fitness center and the third is a home-based version of the program performed at home.
  Arms: 2

SUMMARY:
The purpose of this study is to conduct a 12-month randomized controlled trial comparing the effects of strength training exercise to stretching and relaxation exercise (control) on body composition (bone, muscle and fat mass), energy balance, bone turnover, and physical function (strength, power, gait, balance and self-report physical function and symptoms) in women who experienced premature menopause from chemotherapy for breast cancer.

DETAILED DESCRIPTION:
As a result of treatment, breast cancer survivors typically experience unhealthy changes in body composition (bone, muscle and fat). Treatments disrupt normal bone and energy balance resulting in bone and muscle wasting and fat gain. Premenopausal women are at greatest risk for these declines because most are thrust into early menopause from chemotherapy. Hormone manipulation therapy (i.e., tamoxifen or arimidex) may further affect these tissues. Exercise can prevent bone and muscle loss and promote fat loss. However, the ability of exercise to reverse unfavorable changes in all components of body composition in women experiencing early menopause from breast cancer treatment has not been specifically studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed breast cancer stage I-IIIa
* Completion of a chemotherapy regimen within the previous 5 years
* Premenopausal status (9-12 menstrual cycles/year) at the initiation of chemotherapy
* Complete absence of menstrual cycles for at least 6 months and within one year after starting chemotherapy OR confirmed menopause by blood tests conducted in the last 12 months prior to enrollment.

Exclusion Criteria:

* Presence of any known metastases
* Clinically defined osteoporosis
* Current or previous use of medications known to affect bone metabolism
* Current regular participation (>2x/wk for at least 30 min/session) in planned impact activities (i.e., volleyball, basketball), or resistance training
* A medical condition, disorder, or medication that contraindicates participation in moderate intensity impact or resistance exercise

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (lumbar spine, proximal femur), bone turnover markers (serum osteocalcin, urinary deoxypyridinoline cross-links) muscle mass, fat mass. | 12 months

SECONDARY OUTCOMES:
Maximal muscle strength, leg power, gait, balance, self-report physical function and symptoms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri M Winters, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU School of Nursing, Portland, Oregon, United States

REFERENCES:
- [Result] Winters-Stone KM, Dobek J, Nail LM, Bennett JA, Leo MC, Torgrimson-Ojerio B, Luoh SW, Schwartz A. Impact + resistance training improves bone health and body composition in prematurely menopausal breast cancer survivors: a randomized controlled trial. Osteoporos Int. 2013 May;24(5):1637-46. doi: 10.1007/s00198-012-2143-2. Epub 2012 Sep 21. PMID 22996743
- [Derived] Winters-Stone KM, Wood LJ, Stoyles S, Dieckmann NF. The Effects of Resistance Exercise on Biomarkers of Breast Cancer Prognosis: A Pooled Analysis of Three Randomized Trials. Cancer Epidemiol Biomarkers Prev. 2018 Feb;27(2):146-153. doi: 10.1158/1055-9965.EPI-17-0766. Epub 2017 Nov 15. PMID 29141853